CLINICAL TRIAL: NCT05162430
Title: Inhibitory Effect of Different Doses of Propofol on Perineal Pruritus Caused by Dexamethasone Sodium Phosphate in Patients Undergoing Day Surgery
Brief Title: Inhibitory Effect of Propofol on Perineal Pruritus in Patients Undergoing Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Wang wanxia, student, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: wWang
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pruritus Vulvae
MeSH Terms: conditions — Pruritus Vulvae | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- P1 group (Experimental): Administration of 0.1 mg/kg of propofol and 5mg dexamethasone phosphate sodium
  Interventions: Drug: Propofol
- P2 group (Experimental): Administration of 0.2mg/kg of propofol and 5mg dexamethasone phosphate sodium
  Interventions: Drug: Propofol
- P3 group (Experimental): Administration of 0.3mg/kg of propofol and 5mg dexamethasone phosphate sodium
  Interventions: Drug: Propofol
- P4 group (Experimental): Administration of 0.4 mg/kg of propofol and 5mg dexamethasone phosphate sodium
  Interventions: Drug: Propofol
- P5 group (Experimental): Administration of 0.5mg/kg of propofol and 5mg dexamethasone phosphate sodium
  Interventions: Drug: Propofol
- D1 group (No Intervention): Administration of 5mg dexamethasone phosphate sodium

INTERVENTIONS:
Drug: Propofol — 0.1mg/kg, 0.2mg/kg, 0.3mg/kg, 0.4mg, kg, 0.5mg/kg Propofol was injected to five groups of P1, P2, P3, P4 and P5, respectively, and 5mg dexamethasone sodium phosphate was given to groups P1, P2, P3, P4, P5 and D1 after 30s
  Arms: P1 group; P2 group; P3 group; P4 group; P5 group

SUMMARY:
OBJECTIVE: To investigate the inhibitory effect of different doses of propofol on perineal pruritus induced by dexamethasone sodium phosphate injection in women, with a view to providing clinical reference for comfortable clinical care in day surgery.

METHODS: One hundred and fifty patients with ASA classification I or II undergoing elective day surgery were randomly divided into six groups of P1, P2, P3, P4, P5 and D1, with 25 cases in each group. Before administration of dexamethasone, propofol injection 0.1 mg/kg, 0.2 mg/kg, 0.3 mg/kg, 0.4 mg/kg and 0.5 mg/kg were given intravenously in groups P1, P2, P3, P4 and P5, respectively (injection rate was 5 s), followed by 30 s of intravenous dexamethasone sodium phosphate 10 mg in all five groups; 5 ml of saline was given in group D1, and 30 s After that, dexamethasone sodium phosphate injection was given (injection speed was 5s in all five groups). The perineal itching, the onset and duration of itching, the visual analogue score (VAS) of itching, the sleep disorder sedation score (Ramsay score) and the occurrence of adverse reactions were recorded in the five groups.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years old ASA classification I-II grade Body mass index (BMI) 18-30kg/m2

Exclusion Criteria:

Patients with paresthesia or pruritus Drug and alcohol abuse Allergies to lipid drugs and contraindications; corticosteroids are cautious Patients Hyperlipidemia Patients during pregnancy and lactation Mental diseases, communication disorders Patients who use hormones for a long time

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Duration of pruritus | 3-6 minutes
  After the administration of dexamethasone sodium phosphate, if pruritus occurs, record the beginning and end
Incidence of pruritus | 3-6 minutes
  Calculation of the occurrence of pruritus in each group.
Severity of pruritus | 3-6 minutes
  Pruritus is classified as mild to moderate to severe according to the VAS score.
VAS score | 10-30 seconds
  Patients rate their pruritus according to the VAS scale.
Ramsay score | 10-30 seconds
  Scoring of patients according to their mental status after administration of propofol.

SECONDARY OUTCOMES:
Adverse reactions | 3-6 minutes
  Hypotension, respiratory depression, injection pain after propofol use, record it.

CONTACTS AND LOCATIONS:
Overall Officials: Liu m yu, Director, Principal Investigator — Yangzhou University
Locations (1):
- Liu meiyu, Yangzhou, Jiangsu, China